CLINICAL TRIAL: NCT01177592
Title: Thrombocyte Activity Reassessment and GEnoTyping for PCI(TARGET-PCI)
Acronym: TARGET-PCI
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of financial support
Sponsor: LifeBridge Health (Other)
Responsible Party: Principal Investigator, Kevin Bliden, Sinai Center for Thrombosis Research Program Manager, LifeBridge Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1714
Record Dates: First submitted 2010-08-06; First posted 2010-08-09 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guided Therapy (Experimental): Subjects on chronic clopidogrel therapy (≥ 5 days maintenance or loading within 4 hours of PCI) will be guided by VerifyNow P2Y12 assay, whereas clopidogrel naïve subjects will be guided by Verigene CYP2C19 genotyping assay. Patients on clopidogrel maintenance and/or in the control group will also be genotyped; conversely, clopidogrel naïve subjects will have VerifyNow testing prior to discharge for additional study analysis. Patients in the guided therapy group that have a measurement of ≥ 230 PRU will be reloaded with 60mg prasugrel and receive standard maintenance dosing. Similarly, clopidogrel naïve subjects that are considered CYP2C19*2 carriers will also be reloaded with 60mg prasugrel and receive standard maintenance dosing
  Interventions: Device: VerifyNow, Verigene
- Standard Therapy (No Intervention): Patients randomized to the control arm will remain on 75mg clopidogrel arm throughout the study.

INTERVENTIONS:
Device: VerifyNow, Verigene — Subjects on chronic clopidogrel will be guided by VerifyNow P2Y12 assay, whereas clopidogrel naïve subjects will be guided by Verigene CYP2C19 genotyping assay. Patients on clopidogrel maintenance and/or in the control group will also be genotyped; conversely, clopidogrel naïve subjects will have VerifyNow testing prior to discharge for additional study analysis. Patients in the guided therapy group that have a measurement of ≥ 230 PRU will be reloaded with 60mg prasugrel and receive standard maintenance dosing. Similarly, clopidogrel naïve subjects that are considered CYP2C19*2 carriers will also be reloaded with 60mg prasugrel and receive standard maintenance dosing (see flow schematic).
  Arms: Guided Therapy

SUMMARY:
This is a prospective, single-center, randomized trial including 1500 subjects requiring PCI. Subjects with ischemic heart disease due to stenotic lesions in either native coronary arteries or coronary artery bypass undergoing PCI with stent placement and no contraindication to prolonged dual antiplatelet therapy (≥1 year) are eligible to be in the study. Subjects will be randomized to either guided antiplatelet therapy arm (n=750) or standard therapy arm (n=750) and undergo laboratory testing, antiplatelet adjustment, and clinical follow-up for 1 year.

Patients (non-emergent) presenting for PCI will receive standard pre-procedural PCI care as outlined by the current ACC/AHA guidelines. Subjects will be consented peri- PCI (prior to or within 24 hours of PCI) and then randomized (1:1 ratio) to guide or standard non-guided (control) antiplatelet therapy. Physicians will be blinded to genotyping and platelet function results for subjects randomized to the standard therapy group for the duration of the study or if endpoint is met. Subjects on chronic clopidogrel or prasugrel therapy (≥ 2 weeks) will be guided by VerifyNow P2Y12 assay, whereas clopidogrel naïve subjects will be guided by Verigene CYP2C19 genotyping assay. Patients on clopidogrel maintenance and/or in the control group will also be genotyped; conversely, clopidogrel naïve subjects will have VerifyNow testing prior to discharge for additional study analysis. Patients in the guided therapy group that have a measurement of ≥ 230 PRU will be reloaded with 60mg prasugrel and receive standard maintenance dosing. Similarly, clopidogrel naïve subjects that are considered CYP2C19*2 carriers will also be reloaded with 60mg prasugrel and receive standard maintenance dosing (see flow schematic). Patients randomized to the control arm will remain on 75mg clopidogrel arm throughout the study. All patients will remain on 325mg ASA for one month and 81-162 mg daily ASA thereafter.

Clinical follow-up (office visit) and post-PCI VerifyNow maintenance testing will occur at 2 weeks, 3 months, and 6 months for patients in the guided therapy group. VerifyNow testing, adverse event occurrence and drug compliance will be performed as part of follow-up. Patients having a measurement of ≥ 230 PRU at 2 weeks or the 3 month visit will be reloaded with 60 mg prasugrel and receive standard maintenance dosing thereafter until the 6-month visit. Patients in guided and control study arms will return at 6 months for clinical follow-up and VerifyNow testing. After completing 6 months of the study treatment period, further antiplatelet therapy will be at the physician's discretion. At 1 year, study subjects will be contacted via phone for clinical assessment and antiplatelet compliance. Physicians adjudicating events will be blinded to the therapy assignment.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between ages 18-85.
* Patients undergoing PCI.
* Patients undergoing coronary angiography and possible PCI with planned use of at least one drug-eluting stent (DES). One or more bare metal stents (BMS) may be implanted, and other lesions may be treated without stenting, as long as at least one DES is implanted. However the procedure must be successful and uncomplicated for all lesions (DES + BMS + non stent).
* Indication for the procedure may be stable angina or ischemia, unstable angina, non-ST elevation MI (NSTEMI).
* Have the ability to understand the requirements of the study, including consent for use and disclosure of research-related health information.
* Have the ability to comply with study procedures and protocol, including required study visits.
* A female patient is eligible to enter the study if she is (1) of child-bearing potential and not pregnant or nursing; (2) not of child bearing potential (i.e. has had a hysterectomy, have both ovaries removed, has tubal ligation, or if she is post-menopausal, defined as 24 months without menses).

Exclusion Criteria:

* Cardiovascular

  * Cardiogenic shock.
  * Ischemic Stroke within 6 weeks
  * Planned staged PCI in the next 6 months post-procedure
  * Unsuccessful PCI (post-procedure diameter stenosis >30% with less than TIMI-3 flow in any treated vessel).
  * Patients with in-hospital STEMI confirmed by ECG prior to randomization or those whom require a target vessel revascularization of the index lesion prior to randomization.
  * Major complication during or after PCI such as but not limited to need for balloon pump, acute stent thrombosis, and major bleed.
* Prior or concomitant therapy

  * Concurrent or planned treatment with warfarin.
  * IIb/IIIa Inhibitors within 72 hrs of PCI
  * Current or planned treatment with Cilostazol
  * Current treatment with Prasugrel
* Hemorrhagic risk

  * History of bleeding diathesis or evidence of active abnormal bleeding within 30 days of randomization.
  * History of hemorrhagic stroke or sub-arachnoid hemorrhage at any time or stroke or TIA of any etiology within 30 days of randomization.
  * Major surgery within 6 weeks prior to randomization.
  * Known platelet count of <100,000/mm3.
  * PT > 1.5 x control.
  * HCT < 25% or > 52%.
  * History of gastro-intestinal bleeding within 6 months.
  * Considered by investigator to be at high-risk for bleeding on long-terms clopidogrel therapy.
  * Minor surgical procedures that require cessation of dual antiplatelet therapy and result in significant bleeding are NOT eligible.
* General

  * Known allergy or contraindication to heparin, aspirin, clopidogrel, or prasugrel.
  * Participation in a study of experimental therapy or device within prior 30 days.
  * Creatinine level of greater than 4.0 mg/dl.
  * Known history of alcohol or drug abuse.
  * Pregnant women or women of child-bearing potential not using an acceptable method of contraception.
  * Severe allergy to stainless steel, contrast dye, unfractionated heparin, low molecular weight heparin, or bivalirudin that cannot be adequately pre-medicated.
  * Current enrollment in an investigational drug or device study that has not reached the time period of the primary endpoint.
  * Patients unwilling or unable to complete clinical follow-up for the duration of the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
MACE | 6 months
  To demonstrate a 30% relative risk reduction in post-PCI ischemic event occurrence (composite of cardiovascular death, ischemic stroke, non-fatal myocardial infarction, urgent target vessel revascularization) with personalized guided antiplatelet treatment as compared to standard post-intervention treatment

SECONDARY OUTCOMES:
Major, Minor, and Nuisance Bleeding | 6 months
  To demonstrate no significant differences in major, minor, and nuisance bleeding with guided therapy as compared to conventional therapy.
MACE | 6 months
  To compare CYP2C19 guided therapy with VerifyNow P2Y12 guided approach in relation to MACE.
Predicting MACE | 6 months
  To determine if a combined (genetic and platelet) approach for guiding therapy is superior to a single approach (genetic or platelet) for predicting MACE.
Overcoming HPR | 6 months
  To demonstrate efficacy of prasugrel in overcoming high platelet reactivity as compared to clopidogrel maintenance therapy.
Platelet Reactivity, Verify Now | 6 months
  To determine the stability of platelet reactivity over time as measured by VerifyNow.
VerifyNow and Bleeding | 6 months
  To determine a relation between VerifyNow P2Y12 results and bleeding events (medically relevant major, minor, and nuisance).
Verify Now and Ischemic Event | 6 months
  To determine a relation between VerifyNow P2Y12 results and ischemic event occurrence.
CYP2C19, ischemia and bleeding | 6 months
  To determine the relation of CYP2C19 variants to ischemia and bleeding.
HPR in prasugrel treatment | 6 months
  To determine the incidence of HPR (as define by PRU ≥230) in prasugrel treated subjects.
Genotype guided therapy | 6 months
  To demonstrate feasibility of genotype guided therapy with the Verigene System by evaluation of test turnaround time, ease of use and reliability in a point of care setting.
Algorithm | 6 months
  To develop an optimal or "recommended" algorithm for guided antiplatelet therapy integrating genotyping and platelet function testing.
Utilizing Patient Questionnaire | 6 months
  To assess the utility of the personalized antiplatelet approach in clinical practice (utilizing a physician questionnaire)
Cutpoints for Plateletworks | 6 months
  To determine cutpoints for ischemic and bleeding risk using the Plateletworks Assay.
Platelet Mapping | 6 months
  To determine a relation between platelet mapping results and bleeding.
Platelet Mapping and Ischemic Event | 6 months
  To determine a relation between platelet mapping results and ischemic event occurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Gurbel, M.D., Principal Investigator — Sinai Hospital of Baltimore
Locations (1):
- Sinai Center for Thrombosis Research, Baltimore, Maryland, United States